CLINICAL TRIAL: NCT05803044
Title: Medico Legal Importance of Drug Abuse Detection Before Emergency Operation
Brief Title: Importance of Drug User Detection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wafaa Sadek Tolba, Demonstrator, Assiut University
Other Study IDs: Drug users detection
Record Dates: First submitted 2023-02-03; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Drug Addiction
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Identify the illicit drugs (morphine, cannabinoids, benzodiazepines, barbiturates, tramadol, cocaine, amphetamine, alcohol, synthetic cannabinoids).
2. Identify illicit drug users in patients who admitted in Assiut University Hospitals undergoing emergency operation and their percent among all patients admitted for emergency operation, for proper selection of anaesthetic agents and proper care before, during and after operations.
3. Compare between addict and non addict in using suitable anaesthetic agents and doses - period of anaesthesia- period of recovery- complications.
4. Compare between addict and non addict patients in :( vital signs before, during and after operation by using anaesthetic chart).
5. Identify the importance of using drug abuse detection as a routine lab work before urgent operations.

DETAILED DESCRIPTION:
Drug addiction has become a more common problem worldwide. In many countries drug abuse is rapidly increasing among young generations .By taking routine preoperative history, it has been noticed that there is a high percentage of patients who were addicted to different types of drugs. Drug addiction remarkably increases morbidity and mortality among patients. Addiction could be defined as a chronic disorder characterized by the compulsive use of a substance, resulting in physical, psychological or social harm to the user and continued use despite that harm .

Substances that could be abused are so many: alcohol, sedative and hypnotics, opioids, cocaine and amphetamines, cannabis, hallucinogens and nicotine. They can be classified as socially acceptable drug (e.g., alcohol, tobacco), a medically prescribed drug (e.g., diazepam), and illegal substance (e.g., cocaine) .

Both acute intoxication and chronic abuse of these substances present challenges for anesthetic management during and after an operation .Whereas some procedures may be delayed while the issue is addressed, others are urgent or emergent and the surgeon and anesthesiologist must be able to deal with the physiologic changes that may occur in these patients.

So, it is important to understand the situations of drug users, such as the category of drugs used, the dosage, the duration of drug use, their history of detoxification or abstention, and especially their current abuse of drugs. Pain threshold in addicts is lower than ordinary people who are not addict to opium due to several reasons including change in function, sensitivity reduction, or decrease in opioid's receptors.

Nevertheless, they are more resistant against narcotics and analgesic drugs. With little information about the history of drug abuse, a quick screening for recent use of drugs is important for both medical staff and patients. The immune colloidal gold (ICG) technique is a well-established technique and is commonly used for screening for drug abuse .

Awareness of the drug's pharmacodynamics, pharmacokinetics and interaction with anesthetics medication is crucial to the proper management of illicit drug users during the perioperative period. Moreover, it is common for illicit drug users to have infection with human immune-deficiency virus (HIV), hepatic C virus (HCV), syphilis or other sexually transmitted disease (STD), which may put medical staff in danger. Incidences of intraoperative and postoperative complications are increased in illicit drug users such as pulmonary infection and coagulation disorders .

Death of drug abusers during anaesthesia and intra operative may occur due to severe cardiovascular cocaine toxicity if general stabilization and hemodynamic control not achieved .

The preventable perioperative complications are evaluated to improve the safety of health care, including also the medical-law point of view .

On the other side, research was done in 2016 at Johans Hopkins found that the average of 250.000 people die in US because of medical errors each year. Updating for this study in 2020 found that the serious medical errors occur most frequently in ICU, emergency departments and operation rooms. Many lawsuits are filled each year against doctors.

For these reasons and more it is important, to the patients and medical staff, to make preoperative drug abuse analysis as a mandatory before emergency surgeries to achieve optimal management during and after operations.

ELIGIBILITY:
Inclusion Criteria:

* Emergency operations.
* Age group more than 18 years.

Exclusion Criteria:

* -Age group less than 18 years.
* Patients refuse to be included in the study

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two hundred patients who undergoing emergency operation of both sexes, in age group more than 18 years will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
By using an anaesthetic record sheat | basline
  which will include
  * physiological parameter as:
  * age (years)
  * weight (kg)
  * blood pressure(mmHg)
  * heart rate(beat /min)
  * respiratory rate(breath/ min)

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Mohamed Almaz, lecturer, Study Director — Supervision; Shimaa Abass Hassan, Lecturer, Study Director — Supervision

REFERENCES:
- [Background] Li J, Ma H, Liao R, Huang Y, Chen G. Preoperative screening for illicit drug use in patients undergoing emergency surgery: A prospective observational study. Sci Rep. 2018 May 9;8(1):7405. doi: 10.1038/s41598-018-25829-3. PMID 29743682
- [Background] Mansourian A, Askarzadeh M, Shabani M, Divsalar K. Comparison of Duration of Spinal Anesthesia with Lidocaine or Lidocaine plus Epinephrine between Addicts and Non-addicts. Addict Health. 2012 Summer-Autumn;4(3-4):95-101. PMID 24494142
- See also: Raynes M and Lawn M(2022):shocking medical malpractice statistics for 2021 — http://rayneslaw.com/shocking-medical-malpractice-statistics-for-2021/